CLINICAL TRIAL: NCT06493136
Title: Etude de l'ANesthésie Par Gel de Lidocaïne Pour Les Injections IntrA vitréennes
Acronym: ANGLIA
Status: Completed | Type: Observational
Sponsor: Institut Ophtalmologique de l'Ouest Jules Verne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A00702-41
Record Dates: First submitted 2024-06-25; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Retinal Diseases - AMD - PAIN - Intravitreal Injection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- questionnaire: questionnaire
  Interventions: Drug: lidocaine gel

INTERVENTIONS:
Drug: lidocaine gel — questionnaire

SUMMARY:
Purpose To assess the efficacy of preservative-free Lidocaine gel 2% (LG) in patients complaining of pain during intravitreal injection (IVI) despite standard topical anaesthesia.

Methods First phase: prospective selection of a group of painful patients (score pain ≥ 4 on Visual Analogic Scale) during IVI with anaesthetic drops. Determination of the anxiety score before IVI, the overall pain score and pain score related to the speculum after IVI. Painful patients were proposed to enter the second phase of the study and have the next IVI with LG. Pain scores and anxiety score after each method of anaesthesia were compared.

Results In a group of 240 patients, 62 (25%) described pain≥4 despite anaesthetic drops. 39 patients (16.3%), accepted anaesthesia with LG for the next IVI. During IVI with LG, 27 patients (69%) had pain<4 (P<0.001). The average pain score for IVI with LG was 3.32+/-2.45 versus 5.71 +/-1.45 for anaesthetic drops (P<0.001). Pain score due to speculum placement was 1.54+/-1.96 for LG versus 2.66+/-2.57 for drops (P=0.02). Anxiety score before IVI was 8.08+/-3.63 for LG versus 7.84+/-3.84 with drops (P=0.4). 27 patients (69%) wanted to have subsequent IVIs with LG.

Conclusion In a selected group of painful patients, anaesthesia with Lidocaine gel provided a statistically significant decrease of the pain score during IVI and the speculum placement pain score. The similarity of anxiety score before each method of anaesthesia, suggests that the reduction of pain score was truly due to a superior anaesthetic effect of LG.

DETAILED DESCRIPTION:
Introduction Déterminer l'efficacité d'une anesthésie topique par gel de Lidocaine à 2% (GL) à la place de l'oxybuprocaine chez les patients se plaignant d'une douleur importante lors des injections intravitréennes. (IVT) avec une aiguille 30 gauge.

Matériels et Méthodes Première phase: réalisation d'un premier interrogatoire parmi des patients ayant des IVT unilatérales réalisées par six praticiens pour déterminer 1) la douleur après IVT avec ovybuprocaine, 2) la douleur liée au blépharostat et 3) l'anxiété avant IVT par l'Hospital Anxiety and Depression Scale , et sélectionner un groupe de patients se plaignant d'une douleur ≥ 4 sur une échelle visuelle analogique (EVA) de la douleur et acceptant aussi une anesthésie par GL lors de la prochaine IVT (groupe étudié). Deuxième phase : réalisation d'un deuxième interrogatoire sur le groupe étudié pour déterminer la douleur ressentie après GL (critère principal), déterminer l'anxiété avant les IVT et la douleur lors de la pose du blépharostat. (critères secondaires).

Résultats Sur un groupe de 240 patients 62 (25%) ont décrit une douleur ≥ 4. 39 patients (16,3%) dont 32 femmes (82%) - Age moyen 77 ans ont accepté une anesthésie par GL et ont constitué le groupe étudié. Après IVT avec GL 27 patients (70%) avaient une douleur < 4 (P< 0,001). Le score moyen de douleur après IVT était de 5,71 +/- 1,45 pour l'oxyburpocaine contre 3,32 +/- 2,45 pour le GL (P< 0,001). Lors de la pose du blépharostat la douleur était de 2,66 +/- 2,57 avec l'oxybuprocaine contre 1,54 +/- 1,96 avec le GL (P= 0,02). Le score d'anxiété avant IVT était de 7,84 +/- 3,84 avant IVT avec oxybuprocaine contre 8,08 +/- 3,63 (P=0,4). 27 patients (69%) souhaitaient avoir des IVT ultérieures avec du GL.

Discussion Le gel de Lidocaine possède une autorisation de mise sur le marché pour la chirurgie ophtalmologique. Dans notre étude, il a permis une réduction significative du score de douleur après IVT en comparaison avec une anesthésie précédente par oxybuprocaine. Il a aussi permis une réduction de la douleur lors de la pose du blépharostat. Ce médicament est pour l'instant réservé à un usage professionnel et n'est pas disponible en officine ce qui restreint son utilisation aux IVT réalisées dans des établissements de santé.

Conclusion L'utilisation de Gel de Lidocaine a permis une réduction significative de la douleur après IVT chez un groupe de patients algiques et plus des deux tiers d'entre eux souhaitaient poursuivre les IVT avec ce type d'anesthésique.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a VAS score during the 1st assessment: VAS ≥ 4/10
* Patients who have given their consent to switch to the protocol with the addition of lidocaine gel (information letter provided and collection of non-objection)

Exclusion Criteria:

* Persons cited in articles L.1121-6 to L.1121-8 of the CSP
* Patients not followed at the IOO Jules Verne or at the Hauts Pavés practice.
* Eye pain before the procedure
* Intravitreal injections performed with oftriamcinolone acetonide
* Intravitreal injections performed with a larger gauge needle (Ozurdex® or Iluvien ®)
* Intravitreal injections performed using a disinfectant other than povidone iodine
* Patients for whom the protocol with lidocaine gel in anesthesia is already used
* Any cortisone injection
* Any uveitic inflammatory pathology whether immunological or infectious
* Anyone under systemic treatment with cortisone or morphine and its derivatives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who made an appointment for an Intra Vitreous Injection (IVT) at the IOO Jules Verne during the recruitment period.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale : pain score | 5 minutes after IVT
  VAS score: The figure should be rounded to the nearest millimetre. Comparison of the pain felt during the injection during the 1st evaluation (with conventional anaesthesia) to the pain score pain score obtained with improved anaesthesia.

SECONDARY OUTCOMES:
Pain score on simple verbal scale | 5 minutes after IVT
  Confirmation of pain relief with the simple verbal scale score
Hospital Anxiety and Depression Scale - Auteurs : A.S. Zigmond et R.P. Snaith | Before the IVT
  Description of the patient's psychological state during an iVT and validation of score stability

CONTACTS AND LOCATIONS:
Overall Officials: Jean François DR Le Rouic, DOCTOR, Principal Investigator — Clinique Jules Verne
Locations (1):
- Institut Ophtalmologique de l'Ouest Jules Verne, Nantes, Loire Atlantique, France

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT06493136/Prot_SAP_000.pdf